CLINICAL TRIAL: NCT04048616
Title: Impact of Protein and Alkali Supplementation on Skeletal Muscle in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lisa Ceglia, Associate Professor of Medicine, Tufts University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3010; 1R01AG055443-01A1 (NIH)
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Age-Related Sarcopenia; Muscle Loss
MeSH Terms: conditions — Muscular Atrophy | interventions — potassium bicarbonate; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: double blind randomized placebo controlled 2x2 factorial design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- whey protein isolate + KHCO3 (Active Comparator): 1.5 gm/kg/day of whey protein and 81 mmol/day of KHCO3
  Interventions: Dietary Supplement: whey protein isolate; Dietary Supplement: potassium bicarbonate (KHCO3)
- whey protein isolate + microcrystalline cellulose (Active Comparator): 1.5 gm/kg/day of whey protein and identical placebo microcrystalline cellulose capsules
  Interventions: Dietary Supplement: whey protein isolate; Other: microcrystalline cellulose
- maltodextrin powder + KHCO3 (Active Comparator): isocaloric placebo maltodextrin powder and 81 mmol/day of KHCO3
  Interventions: Dietary Supplement: potassium bicarbonate (KHCO3); Other: maltodextrin powder
- maltodextrin powder + microcrystalline cellulose (Placebo Comparator): isocaloric placebo maltodextrin powder and identical placebo microcrystalline cellulose capsules
  Interventions: Other: microcrystalline cellulose; Other: maltodextrin powder

INTERVENTIONS:
Dietary Supplement: whey protein isolate — one 15-25 gm (based on body weight) protein packet three times a day with each meal
  Arms: whey protein isolate + KHCO3; whey protein isolate + microcrystalline cellulose
Dietary Supplement: potassium bicarbonate (KHCO3) — two 13.5 mmol capsules three times a day with each meal
  Arms: maltodextrin powder + KHCO3; whey protein isolate + KHCO3
Other: microcrystalline cellulose — identical placebo capsule
  Arms: maltodextrin powder + microcrystalline cellulose; whey protein isolate + microcrystalline cellulose
Other: maltodextrin powder — isocaloric placebo powder
  Arms: maltodextrin powder + KHCO3; maltodextrin powder + microcrystalline cellulose

SUMMARY:
The central hypothesis is that higher protein intake and a neutralizing alkaline salt supplement will improve muscle performance and mass, compared to their respective placebos, in older men and postmenopausal women.

DETAILED DESCRIPTION:
With aging, skeletal muscle mass and performance decline leading to an increased risk of falls and physical disability. There is ongoing research on whether increasing dietary protein intake in older adults improves indices of muscle health and thus translates to a reduction in physical disability. A main concern is that high protein results in a large dietary acid load from the breakdown of protein to acidogenic byproducts, which could in turn promote muscle degradation particularly in older adults with age-related declines in renal excretion of acid. The scientific premise of this project is that the balance between the amount of protein in the diet (anabolic component) and the net acid load of the diet (catabolic component) in part determines whether the diet as a whole has a net anabolic or catabolic effect on muscle. Preliminary data have suggested that a daily alkaline salt supplement (potassium bicarbonate, KHCO3) lowered the dietary acid load and improved lower extremity muscle power in postmenopausal women.

The investigator's central hypothesis is that higher protein intake and a neutralizing alkaline salt will improve muscle performance and mass, compared to their respective placebos, in older men and postmenopausal women. To test the hypothesis, the investigators conducted a randomized, double-blind, placebo-controlled, 2x2 factorial study in underactive men and women age 65 and older on baseline lower protein diets. Participants were assigned to one of four groups: either a whey protein supplement (to raise protein intake to 1.5 g/kg/d) with or without KHCO3 81 mmol/d or an isocaloric placebo supplement with or without KHCO3 81 mmol/d for 24 wks.

ELIGIBILITY:
Inclusion Criteria:

1. ability to sign informed consent form
2. ambulatory community-dwelling men and women
3. age 65 years and over
4. habitual dietary intake of protein of ≤0.8 g/kg/d
5. underactive
6. estimated glomerular filtration rate ≥ 50 ml/min/1.73 m2

Exclusion Criteria:

1. participation in a diet or intensive exercise program during the study
2. vegetarian (no animal protein)
3. oral glucocorticoid use for > 10 days in the last 3 months
4. anabolic and gonadal hormones in the last 6 months
5. Tamoxifen/raloxifene in the last 6 months
6. regular use of alkali-producing antacids (> 3 times per week)
7. potassium-containing supplements or products
8. non-steroidal anti-inflammatory medications >3 times per week
9. antacids containing calcium carbonate, aluminum hydroxide, magnesium hydroxide, or calcium acetate
10. insulin
11. sulfonylureas
12. SGLT2 inhibitors
13. a lower extremity fracture in the last year
14. kidney stones in the past 5 years
15. hyperkalemia
16. elevated serum bicarbonate
17. hypercalcemia
18. uncontrolled diabetes mellitus defined as having fasting blood >150 or hemoglobin A1c >8%
19. untreated thyroid or parathyroid disease
20. significant immune disorder
21. current unstable heart disease
22. Crohn's disease
23. active malignancy or cancer therapy in the last year
24. alcohol use exceeding 2 drinks/day
25. current peptic ulcers or esophageal stricture
26. other condition or abnormality in screening labs, at discretion of the study physician

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 141 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Ceglia, MD MS, Principal Investigator — Tufts Medical Center and Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2021 to July 2023, ambulatory, community-dwelling men and postmenopausal women aged 65 years and older were recruited from direct mailings to the HNRCA volunteer database and the Tufts Medical Center patient database.
Pre-assignment Details: Exclusion criteria included use of oral glucocorticoids, anabolic and gonadal hormones, alkali-producing antacids, potassium-containing supplements, insulin, uncontrolled diabetes mellitus, kidney stones, advanced chronic kidney disease, cirrhosis, gastroesophageal or intestinal disease, immune disorders, unstable heart disease, untreated thyroid or parathyroid disease, active malignancy or cancer therapy, recent fracture, milk protein allergy, and relevant laboratory abnormalities.
Period: Overall Study
Arm/Group | Whey Protein Isolate + KHCO3 | Whey Protein Isolate + Microcrystalline Cellulose | Maltodextrin Powder + KHCO3 | Maltodextrin Powder + Microcrystalline Cellulose
Started | 35 | 36 | 35 | 35
Completed | 29 | 32 | 31 | 31
Not Completed | 6 | 4 | 4 | 4

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat sample of 128 participants with available outcome data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Whey Protein Isolate + KHCO3 | Whey Protein Isolate + Microcrystalline Cellulose | Maltodextrin Powder + KHCO3 | Maltodextrin Powder + Microcrystalline Cellulose | Total
Number analyzed (Participants) | 29 | 34 | 31 | 34 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 29 | 34 | 31 | 34 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.1 (6.4) | 74.5 (6.3) | 74.1 (5.3) | 72.7 (5.5) | 74.1 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 16 | 16 | 61
  Male | 15 | 19 | 15 | 18 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 28 | 34 | 31 | 33 | 126
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 4 | 0 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 3 | 1 | 4 | 5 | 13
  White | 25 | 29 | 25 | 28 | 107
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 34 | 31 | 34 | 128

OUTCOME MEASURES:

1. Primary Outcome: Double Leg Press Peak Power at 70%
Description: Double leg press peak power at 70% of the 1 repetition maximum
Time Frame: 24 weeks
Population: Analysis used an at-the-margins approach to evaluate the superiority of whey protein (WP) against placebo-WP and of potassium bicarbonate (KHCO3) against placebo-KHCO3
Measure: Mean (95% Confidence Interval); unit: Watts
Groups:
- Whey Protein (WP): Combined participants assigned to the WP + potassium bicarbonate (KHCO3) group and the WP + microcrystalline cellulose placebo
- Placebo-WP: Combined participants assigned to the maltodextrin + KHCO3 group and the maltodextrin + microcrystalline cellulose placebo group
- Potassium Bicarbonate (KHCO3): Combined participants assigned to the KHCO3 + WP group and the KHCO3 + maltodextrin placebo
- Placebo-KHCO3: Combined participants assigned to the microcrystalline cellulose placebo + WP group and the microcrystalline cellulose placebo + maltodextrin placebo group
Arm/Group | Whey Protein (WP) | Placebo-WP | Potassium Bicarbonate (KHCO3) | Placebo-KHCO3
Number analyzed (Participants) | 59 | 61 | 60 | 60
Watts | 260.3 [241.9 to 278.7] | 255.6 [237.5 to 273.7] | 251.1 [232.9 to 269.3] | 264.8 [246.4 to 283.1]

2. Secondary Outcome: Double Leg Press Peak Power at 70%
Description: Double leg press peak power at 70% of the 1-repetition maximum
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Watts
Arm/Group | Whey Protein (WP) | Placebo-WP | Potassium Bicarbonate (KHCO3) | Placebo-KHCO3
Number analyzed (Participants) | 60 | 62 | 59 | 63
Watts | 252.8 [233.4 to 272.2] | 253.8 [234.8 to 272.8] | 246.9 [227.4 to 266.4] | 259.7 [240.8 to 278.7]

3. Secondary Outcome: Double Leg Press Peak Power at 40%
Description: Double leg press peak power at 40% of the 1 repetition maximum
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Watts
Arm/Group | Whey Protein (WP) | Placebo-WP | Potassium Bicarbonate (KHCO3) | Placebo-KHCO3
Number analyzed (Participants) | 59 | 61 | 60 | 63
Watts | 223.8 [200.4 to 247.3] | 219.5 [196.5 to 242.6] | 225.3 [202.0 to 248.5] | 218.1 [194.6 to 241.5]

4. Secondary Outcome: Double Leg Press Peak Power at 40%
Description: Double leg press peak power at 40% of the 1 repetition maximum
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Watts
Arm/Group | Whey Protein (WP) | Placebo-WP | Potassium Bicarbonate (KHCO3) | Placebo-KHCO3
Number analyzed (Participants) | 60 | 63 | 60 | 63
Watts | 221.9 [199.5 to 244.3] | 215.8 [193.8 to 237.7] | 220.7 [188.3 to 253.1] | 215.3 [192.7 to 237.8]

5. Secondary Outcome: Knee Extension Peak Torque
Description: Knee extension peak torque at 60 degrees/s using Biodex Isokinetic Dynamometer
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Newton-meters
Arm/Group | Whey Protein (WP) | Placebo-WP | Potassium Bicarbonate (KHCO3) | Placebo-KHCO3
Number analyzed (Participants) | 61 | 62 | 60 | 63
Newton-meters | 99.5 [95.6 to 103.3] | 101.5 [97.7 to 105.3] | 102.4 [98.5 to 106.2] | 98.6 [94.8 to 102.4]

6. Secondary Outcome: Knee Extension Peak Torque
Description: Knee extension peak torque at 60 degrees/s using Biodex Isokinetic Dynamometer
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: Newton-meters
Arm/Group | Whey Protein (WP) | Placebo-WP | Potassium Bicarbonate (KHCO3) | Placebo-KHCO3
Number analyzed (Participants) | 63 | 65 | 60 | 68
Newton-meters | 96.2 [92.6 to 99.8] | 100.8 [97.4 to 104.3] | 95.2 [87.2 to 103.2] | 97.7 [94.1 to 101.3]

7. Secondary Outcome: Handgrip Strength
Description: Measure maximum handgrip strength in either hand using handheld Jamar+ dynamometer
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Whey Protein (WP) | Placebo-WP | Potassium Bicarbonate (KHCO3) | Placebo-KHCO3
Number analyzed (Participants) | 61 | 62 | 60 | 63
kg | 29.0 [27.8 to 30.1] | 28.3 [27.2 to 29.4] | 28.7 [26.7 to 29.8] | 28.5 [27.4 to 29.6]

8. Secondary Outcome: Appendicular Lean Body Mass/Height Squared
Description: Dual energy X-ray absorptiometry (DXA) lean mass of arms plus legs divided by height squared
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Whey Protein (WP) | Placebo-WP | Potassium Bicarbonate (KHCO3) | Placebo-KHCO3
Number analyzed (Participants) | 60 | 62 | 60 | 62
kg/m^2 | 7.0 [6.9 to 7.1] | 7.1 [7.0 to 7.1] | 7.0 [6.9 to 7.1] | 7.1 [7.0 to 7.2]

9. Secondary Outcome: Physical Performance Battery Score
Description: Performance score (range 0-4 with higher values representing a better performance) based on Health Aging and Body Composition-Physical Performance Battery
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Whey Protein (WP) | Placebo-WP | Potassium Bicarbonate (KHCO3) | Placebo-KHCO3
Number analyzed (Participants) | 61 | 62 | 60 | 63
score on a scale | 2.1 [2.0 to 2.2] | 2.2 [2.1 to 2.3] | 2.2 [2.1 to 2.3] | 2.1 [2.1 to 2.2]

10. Secondary Outcome: 24 Hour Urinary Total Nitrogen Excretion
Description: Measure based on 24 hour urine total nitrogen excretion
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: g
Arm/Group | Whey Protein (WP) | Placebo-WP | Potassium Bicarbonate (KHCO3) | Placebo-KHCO3
Number analyzed (Participants) | 61 | 63 | 60 | 63
g | 13.1 [12.2 to 14.0] | 9.8 [8.9 to 10.7] | 11.2 [10.3 to 12.1] | 11.7 [10.9 to 12.6]

11. Other Pre Specified Outcome: D3-creatine Muscle Mass/Weight
Description: measure of total body percent muscle mass by D3-creatine dilution method
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of muscle mass
Arm/Group | Whey Protein (WP) | Placebo-WP | Potassium Bicarbonate (KHCO3) | Placebo-KHCO3
Number analyzed (Participants) | 57 | 58 | 55 | 60
percentage of muscle mass | 27.9 [27.1 to 28.8] | 29.1 [28.3 to 29.9] | 28.9 [28.1 to 29.7] | 28.1 [27.3 to 29.0]

12. Post Hoc Outcome: IGF-1
Description: Serum insulin-like growth factor 1 (IGF-1) level
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Whey Protein (WP) | Placebo-WP | Potassium Bicarbonate (KHCO3) | Placebo-KHCO3
Number analyzed (Participants) | 61 | 61 | 59 | 63
ng/mL | 118.5 [113.8 to 123.3] | 104.3 [99.6 to 109.0] | 115.0 [110.2 to 119.8] | 107.8 [103.2 to 112.5]

ADVERSE EVENTS:
Time Frame: up to 24 weeks
Description: Standard definitions
Arm/Group | Whey Protein Isolate + KHCO3 | Whey Protein Isolate + Microcrystalline Cellulose | Maltodextrin Powder + KHCO3 | Maltodextrin Powder + Microcrystalline Cellulose
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36 | 0/35 | 1/35
Serious Adverse Events (participants affected / at risk) | 3/35 | 2/36 | 3/35 | 3/35
Other Adverse Events (participants affected / at risk) | 22/35 | 14/36 | 18/35 | 14/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Whey Protein Isolate + KHCO3 (N=35) | Whey Protein Isolate + Microcrystalline Cellulose (N=36) | Maltodextrin Powder + KHCO3 (N=35) | Maltodextrin Powder + Microcrystalline Cellulose (N=35)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cardiovascular event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Fall with musculoskeletal complication (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Whey Protein Isolate + KHCO3 (N=35) | Whey Protein Isolate + Microcrystalline Cellulose (N=36) | Maltodextrin Powder + KHCO3 (N=35) | Maltodextrin Powder + Microcrystalline Cellulose (N=35)
Pedal edema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myocardial infaction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
coronary heart disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign Positional Vertgo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 3 (3) | 5 (6) | 3 (3)
Respiratory infections (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4) | 5 (5) | 3 (3)
GERD (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall with injury (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Leg cramps (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Basal cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate problems (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cerebrovascular event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dental infection (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lightheadedness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT04048616/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT04048616/SAP_001.pdf